CLINICAL TRIAL: NCT02472886
Title: A Phase 3b, Multicenter, Open-Label Study to Evaluate the Safety and Efficacy of Ledipasvir/Sofosbuvir in Adults With Chronic HCV Infection
Brief Title: Safety and Efficacy of Ledipasvir/Sofosbuvir in Adults With Chronic HCV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-1463; 2015-000690-13 (EudraCT Number)
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C Virus Infection
Keywords: HCV genotype 1; HCV; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; GS-7977; GS-5885; Ribavirin; Sofosbuvir; ledipasvir; Hepatitis C; Hepatitis C, Chronic; Liver Diseases; Virus Diseases; Antiviral Agents; HCV/HIV co-infection
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic; Liver Diseases; Virus Diseases | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- LDV/SOF (Experimental): Treatment-naive participants with genotype 1 HCV infection without cirrhosis will receive LDV/SOF FDC for 8 weeks.
  Interventions: Drug: LDV/SOF
- LDV/SOF Coinfected with HIV-1 (Experimental): Treatment-naive participants with genotype 1 HCV infection without cirrhosis and who are coinfected with HIV-1 will receive LDV/SOF FDC for 8 weeks.
  Interventions: Drug: LDV/SOF
- LDV/SOF+RBV Retreatment (Experimental): Participants with genotype 1 or 3 HCV infection who failed to achieve SVR12 in Gilead Study GS-US-334-0119 will receive LDV/SOF FDC + RBV for 12 weeks.
  Interventions: Drug: LDV/SOF; Drug: RBV

INTERVENTIONS:
Drug: LDV/SOF — 90/400 mg FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977
Drug: RBV — Tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: LDV/SOF+RBV Retreatment

SUMMARY:
The primary objectives of this study are to evaluate the antiviral efficacy, safety, and tolerability of ledipasvir/sofosbuvir (LDV/SOF) fixed dose combination (FDC) with or without ribavirin (RBV) in adults with chronic hepatitis C virus (HCV) infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants who failed treatment in Study GS-US-334-0119 who meet relevant inclusion/exclusion criteria are eligible for retreatment in this study
* Chronic genotype 1 HCV infection
* HCV treatment-naive
* HCV RNA > 10,000 IU/mL at screening
* Absence of cirrhosis
* Screening laboratory values within defined thresholds
* Use of two effective contraception methods if female of childbearing potential or sexually active male

Key Exclusion Criteria:

* Pregnant or nursing female or male with pregnant female partner
* Infection with hepatitis B virus (HBV)
* Current or prior history of clinical hepatic decompensation
* Chronic use of systemic immunosuppressive agents
* History of clinically significant illness or any other medical disorder that may interfere with the individual's treatment, assessment, or compliance with the protocol
* For HIV-1/HCV co-infected individuals:

  * Opportunistic infection within 6 months prior to screening
  * Active, serious infection (other than HIV-1 or HCV) requiring parental antibiotics, antivirals or antifungals within 30 days prior to baseline
  * Treatment with an antiretroviral (ARV) regimen other than one of those listed in the study protocol

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-06-17 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (9):
- Estonia (2):
  - Tallinn
  - Tartu
- Russia (7):
  - Krasnoyarsk
  - Moscow
  - Saint Petersburg
  - Samara
  - Stavropol
  - Tyumen
  - Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Zhdanov K., Morozov V., Orlova-Morozova E.A., Salupere R., Kozhevnikova G., et al. Preliminary Results of an Evaluation of Ledipasvir/Sofosbuvir in Treatment-Naive Patients with Chronic HCV or HCV/HIV Co-Infection and Retreatment of Sofosbuvir-treated Patients. 8th International Conference of the White Nights of Hepatology. Saint Petersburg, Russia. June 2-3, 2016. Oral presentation.
- [Derived] Isakov V, Gankina N, Morozov V, Kersey K, Lu S, Osinusi A, Svarovskaia E, Brainard DM, Salupere R, Orlova-Morozova E, Zhdanov K. Ledipasvir-Sofosbuvir for 8 Weeks in Non-Cirrhotic Patients with Previously Untreated Genotype 1 HCV Infection +/- HIV-1 Co-Infection. Clin Drug Investig. 2018 Mar;38(3):239-247. doi: 10.1007/s40261-017-0606-0. PMID 29177645

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Russia and Estonia. The first participant was screened on 17 June 2015. The last study visit occurred on 30 June 2016.
Pre-assignment Details: 169 participants were screened.
Groups:
- LDV/SOF 8 Weeks (TN, HCV-monoinfected): Ledipasvir/sofosbuvir (LDV/SOF; Harvoni®) (90/400 mg) fixed dose combination (FDC) tablet once daily for 8 weeks in treatment-naive (TN) participants with genotype 1 HCV infection without cirrhosis
- LDV/SOF 8 Weeks (TN, HCV/HIV-coinfected): LDV/SOF (90/400 mg) FDC tablet once daily for 8 weeks in treatment naive participants with genotype 1 HCV infection without cirrhosis and coinfected with HIV-1
- LDV/SOF + RBV 12 Weeks (TE, SOF-treated, HCV-monoinfected): LDV/SOF (90/400 mg) FDC tablet once daily + weight-based ribavirin (RBV) (1000-1200 mg in a divided daily dose) for 12 weeks in treatment-experienced (TE) participants with genotype 1 or 3 HCV infection who failed to achieve sustained virologic response (SVR) in a previous Gilead sofosbuvir (SOF) study
Period: Overall Study
Arm/Group | LDV/SOF 8 Weeks (TN, HCV-monoinfected) | LDV/SOF 8 Weeks (TN, HCV/HIV-coinfected) | LDV/SOF + RBV 12 Weeks (TE, SOF-treated, HCV-monoinfected)
Started | 67 | 59 | 27
Completed | 67 | 57 | 26
Not Completed | 0 | 2 | 1
Not completed — Lack of Efficacy | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- LDV/SOF 8 Weeks (TN, HCV-monoinfected): LDV/SOF(90/400 mg) FDC tablet once daily for 8 weeks in treatment-naive (TN) participants with genotype 1 HCV infection without cirrhosis
- LDV/SOF + RBV 12 Weeks (TE, SOF-treated, HCV-monoinfected): LDV/SOF (90/400 mg) FDC tablet once daily + weight-based ribavirin (RBV) (1000-1200 mg in a divided daily dose) for 12 weeks in treatment-experienced (TE) participants with genotype 1 or 3 HCV infection who failed to achieve SVR in a previous Gilead sofosbuvir study
- Total: Total of all reporting groups
Arm/Group | LDV/SOF 8 Weeks (TN, HCV-monoinfected) | LDV/SOF 8 Weeks (TN, HCV/HIV-coinfected) | LDV/SOF + RBV 12 Weeks (TE, SOF-treated, HCV-monoinfected) | Total
Number analyzed (Participants) | 67 | 59 | 27 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12.6) | 34 (5.5) | 47 (11.2) | 40 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 25 | 9 | 67
  Male | 34 | 34 | 18 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 66 | 59 | 27 | 152
  Asian | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 67 | 59 | 27 | 153
Region of Enrollment [Count of Participants; unit: Participants]
  Russian Federation | 61 | 47 | 27 | 135
  Estonia | 6 | 12 | 0 | 18
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 17 | 9 | 7 | 33
    CT | 41 | 41 | 18 | 100
    TT | 9 | 9 | 2 | 20
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 5.9 (0.72) | 6.1 (0.54) | 6.3 (0.67) | 6.0 (0.66)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 29 | 23 | 8 | 60
  ≥ 800,000 IU/mL | 38 | 36 | 19 | 93
Cirrhosis Status [Count of Participants; unit: Participants]
  No | 67 | 59 | 17 | 143
  Yes | 0 | 0 | 10 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ) 12 weeks following the last dose of study drug.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set (FAS) included participants who were enrolled into the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- LDV/SOF 8 Weeks (TN, HCV-monoinfected): LDV/SOF (90/400 mg) FDC tablet once daily for 8 weeks in treatment-naive (TN) participants with genotype 1 HCV infection without cirrhosis
Arm/Group | LDV/SOF 8 Weeks (TN, HCV-monoinfected) | LDV/SOF 8 Weeks (TN, HCV/HIV-coinfected) | LDV/SOF + RBV 12 Weeks (TE, SOF-treated, HCV-monoinfected)
Number analyzed (Participants) | 67 | 59 | 27
percentage of participants | 100.0 [94.6 to 100.0] | 96.6 [88.3 to 99.6] | 96.3 [81.0 to 99.9]

2. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to Any Adverse Event (AE)
Time Frame: Up to 12 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Groups:
- LDV/SOF 8 Weeks (TN, HCV-monoinfected): LDV/SOF (90/400 mg) FDC tablet once daily for 8 weeks in treatment-naive participants with genotype 1 HCV infection without cirrhosis
Arm/Group | LDV/SOF 8 Weeks (TN, HCV-monoinfected) | LDV/SOF 8 Weeks (TN, HCV/HIV-coinfected) | LDV/SOF + RBV 12 Weeks (TE, SOF-treated, HCV-monoinfected)
Number analyzed (Participants) | 67 | 59 | 27
percentage of participants | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF 8 Weeks (TN, HCV-monoinfected) | LDV/SOF 8 Weeks (TN, HCV/HIV-coinfected) | LDV/SOF + RBV 12 Weeks (TE, SOF-treated, HCV-monoinfected)
Number analyzed (Participants) | 67 | 59 | 27
percentage of participants
  SVR4 | 100.0 [94.6 to 100.0] | 96.6 [88.3 to 99.6] | 96.3 [81.0 to 99.9]
  SVR24 | 100.0 [94.6 to 100.0] | 96.6 [88.3 to 99.6] | 96.3 [81.0 to 99.9]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ on Treatment
Time Frame: Up to 12 weeks
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF 8 Weeks (TN, HCV-monoinfected) | LDV/SOF 8 Weeks (TN, HCV/HIV-coinfected) | LDV/SOF + RBV 12 Weeks (TE, SOF-treated, HCV-monoinfected)
Number analyzed (Participants) | 67 | 59 | 27
percentage of participants
  Week 1 | 20.9 [11.9 to 32.6] | 39.0 [26.5 to 52.6] | 3.7 [0.1 to 19.0]
  Week 2 | 65.7 [53.1 to 76.8] | 69.5 [56.1 to 80.8] | 59.3 [38.8 to 77.6]
  Week 4 | 100.0 [94.6 to 100.0] | 96.6 [88.3 to 99.6] | 88.9 [70.8 to 97.6]
  Week 8 | 100.0 [94.6 to 100.0] | 98.3 [90.9 to 100.0] | 100.0 [87.2 to 100.0]
  Week 12 | NA [NA to NA] — Treatment for this group was 8 weeks only. | NA [NA to NA] — Treatment for this group was 8 weeks only. | 100.0 [87.2 to 100.0]

5. Secondary Outcome: HCV RNA Change From Day 1
Time Frame: Up to 12 weeks
Population: Participants in Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF 8 Weeks (TN, HCV-monoinfected) | LDV/SOF 8 Weeks (TN, HCV/HIV-coinfected) | LDV/SOF + RBV 12 Weeks (TE, SOF-treated, HCV-monoinfected)
Number analyzed (Participants) | 67 | 59 | 27
log10 IU/mL
  Week 1: number analyzed (Participants) | 65 | 58 | 27
  Week 1 | -3.97 (0.675) | -4.34 (0.626) | -4.12 (0.582)
  Week 2: number analyzed (Participants) | 67 | 58 | 27
  Week 2 | -4.50 (0.687) | -4.76 (0.522) | -4.83 (0.630)
  Week 4 | -4.74 (0.723) | -4.89 (0.534) | -5.08 (0.642)
  Week 8 | -4.74 (0.723) | -4.91 (0.536) | -5.11 (0.671)
  Week 12 | NA (NA) — Treatment for this group was 8 weeks only. | NA (NA) — Treatment for this group was 8 weeks only. | -5.11 (0.671)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as
  * On-treatment virologic failure
    * confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ, while on treatment (ie, breakthrough),
    * confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment (ie, rebound), HCV RNA persistently ≥ LLOQ through 8 weeks of treatment (ie, nonresponse)
  * Relapse
    * HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available posttreatment measurement
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Groups:
- LDV/SOF 8 Weeks (TN, HCV-monoinfected): LDV/SOF (90/400 mg) FDC tablet once daily for 8 weeks in treatment-naive participants with genotype 1 HCV infection without cirrhosiss
Arm/Group | LDV/SOF 8 Weeks (TN, HCV-monoinfected) | LDV/SOF 8 Weeks (TN, HCV/HIV-coinfected) | LDV/SOF + RBV 12 Weeks (TE, SOF-treated, HCV-monoinfected)
Number analyzed (Participants) | 67 | 59 | 27
percentage of participants | 0 | 3.4 | 3.7

7. Secondary Outcome: Percentage of HIV/HCV- Coinfected Participants That Maintain HIV-1 RNA < 50 Copies/mL While on HCV Treatment and at Posttreatment Week 4
Time Frame: Up to Posttreatment Week 4
Population: Participants in the Safety Analysis Set (who had HIV RNA < 50 Copies/mL at baseline) with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 8 Weeks (TN, HCV/HIV-coinfected)
Number analyzed (Participants) | 45
percentage of participants
  Week 4 | 100.0
  Week 8: number analyzed (Participants) | 43
  Week 8 | 100.0
  Posttreatment Week 4: number analyzed (Participants) | 36
  Posttreatment Week 4 | 97.2

8. Secondary Outcome: For HIV/HCV- Coinfected Participants, Change From Baseline in CD4 T-cell Count at the End of Treatment and Posttreatment Week 4
Time Frame: Up to Posttreatment Week 4
Population: Participant in the Safety analysis set (with or without prior antiretroviral (ARV) treatment) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Groups:
- LDV/SOF 8 Weeks (TN, HCV/HIV-coinfected, ARV- Naive): LDV/SOF (90/400 mg) FDC tablet once daily for 8 weeks in treatment naive participants with genotype 1 HCV infection without cirrhosis and coinfected with HIV-1. These participants did not receive any prior ARV therapy.
- LDV/SOF 8 Weeks (TN, HCV/HIV-coinfected, ARV Experienced): LDV/SOF (90/400 mg) FDC tablet once daily for 8 weeks in treatment naive participants with genotype 1 HCV infection without cirrhosis and coinfected with HIV-1. These participants were on a stable ARV regimen for at least 8 weeks prior to screening.
Arm/Group | LDV/SOF 8 Weeks (TN, HCV/HIV-coinfected, ARV- Naive) | LDV/SOF 8 Weeks (TN, HCV/HIV-coinfected, ARV Experienced)
Number analyzed (Participants) | 44 | 9
cells/µL
  Change at Week 4: number analyzed (Participants) | 43 | 9
  Change at Week 4 | 47 (120.5) | 159 (114.9)
  Change at Week 8 | 45 (122.7) | 202 (178.1)
  Change at Posttreatment Week 4: number analyzed (Participants) | 35 | 5
  Change at Posttreatment Week 4 | 74 (117.8) | 172 (114.1)

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | LDV/SOF 8 Weeks (TN, HCV-monoinfected) | LDV/SOF 8 Weeks (TN, HCV/HIV-coinfected) | LDV/SOF + RBV 12 Weeks (TE, SOF-treated, HCV-monoinfected)
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/59 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/59 | 0/27
Other Adverse Events (participants affected / at risk) | 5/67 | 2/59 | 8/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 8 Weeks (TN, HCV-monoinfected) (N=67) | LDV/SOF 8 Weeks (TN, HCV/HIV-coinfected) (N=59) | LDV/SOF + RBV 12 Weeks (TE, SOF-treated, HCV-monoinfected) (N=27)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3
Asthenia (General disorders) | 1 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 2
Headache (Nervous system disorders) | 4 | 0 | 4
Irritability (Psychiatric disorders) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years